CLINICAL TRIAL: NCT05026632
Title: Safety and Efficacy of NPI-002 Intravitreal Implant for the Delay of Cataract Progression in Patients Undergoing Vitrectomy
Brief Title: NPI-002 Intravitreal Implant for the Delay of Cataract Progression
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nacuity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C-21-01
Record Dates: First submitted 2021-08-24; First posted 2021-08-30 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single NPI-002 Intravitreal Implant (Experimental): one NPI-002 implant inserted at the time of vitrectomy
  Interventions: Drug: NPI-002 Intravitreal Implant
- Double NPI-002 Intravitreal Implant (Experimental): two NPI-002 implants inserted at the time of vitrectomy
  Interventions: Drug: NPI-002 Intravitreal Implant
- Control (No Intervention): No implant inserted at time of vitrectomy

INTERVENTIONS:
Drug: NPI-002 Intravitreal Implant — Implant inserted during vitrectomy.
  Arms: Double NPI-002 Intravitreal Implant; Single NPI-002 Intravitreal Implant

SUMMARY:
This study will examine the safety and efficacy NPI-002 intravitreal implants post vitrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Indicated for vitrectomy
2. Natural Lens in place at time of vitrectomy
3. Some cataract present as assessed pre-operatively

Exclusion Criteria:

1. Previous intraocular surgery in study eye.
2. Clear zonular weakness or defects / coloboma.
3. Not on stable dose of medications for other conditions.
4. Need for oral corticosteroids during study participation.
5. Evidence or history of uveitis, or ocular ischemia.
6. Current smoker
7. Use of supplemental oxygen
8. Evidence or history of proliferative diabetic retinopathy.
9. Current lung disease (PU, COPD, Asthma) resulting in decreased oxygen saturation.
10. Sensitivity to thiol compounds.
11. Participation in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-27 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Lens Densitometry | 6 months
  Change from Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jami R Kern, PhD, Study Director — Nacuity Pharmaceuticals
Locations (1):
- Royal Adelaide Hospital, Adelaide, Australia

IPD SHARING:
Plan to Share IPD: No